CLINICAL TRIAL: NCT01064895
Title: Post-Market Observation Study of Intra-renal Drug Delivery (PROVIDE)
Acronym: PROVIDE
Status: Terminated | Type: Observational
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008-CL0015 Revision C
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Acute Kidney Injury; Acute Renal Failure; Renal Failure Chronic Contrast Induced; Chronic Kidney Disease
Keywords: Benephit; Acute Kidney Injury; Acute Renal Failure; Contrast Induced Nephropathy; Chronic Kidney Disease
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Active Cohort: Patients receiving the Benephit device and targeted renal therapy.
  Interventions: Device: Benephit catheter for Targeted Renal Therapy

INTERVENTIONS:
Device: Benephit catheter for Targeted Renal Therapy — Local physician-specified agent delivery to the kidneys bilaterally via the renal arteries using the Benephit infusion system.
  Other Names: Benephit CV,PV,XT Infusion Systems(K033569,K050205,K082163)

SUMMARY:
This is a prospective, observational, multi-center study with consecutive enrollment. Up to 500 patients will be enrolled. All (consecutive) adult patients in whom one or more components of the Benephit Infusion System are planned to be used at participating sites are eligible for enrollment. The objective of this post-marketing surveillance study is to collect clinical usage patterns of the Benephit Infusion Systems. As a result, AngioDynamics will be able to (1) Better understand and quantify usage patterns including patient characteristics, adjunctive procedures, and infusion agents, (2) Collect user-interface information and overall customer satisfaction, and (3) Monitor post-marketing device performance and safety for ISO quality adherence.

DETAILED DESCRIPTION:
Acute kidney injury, or AKI, is a rapid decline in renal function characterized by a decrease in urine output and/or an increase in serum creatinine (Cr), and is associated with worsened clinical outcomes and increased healthcare costs. AKI may be caused by numerous factors including interruptions or perturbations of renal blood flow or toxins, and often these factors are extra-renal in origin. AKI diagnoses in hospitalized patients are over one million per year and are projected to continue to grow, due largely to the aging population and increasing numbers of medical and invasive procedures performed on the elderly and the ever-increasing prevalence of diabetes mellitus and its medical complications, as well as increasing awareness within the medical community.

Treatment options for established acute kidney injury are limited and consist mainly of fluid and electrolyte balance (diuretics and/or IV fluids) supportive care up until the point that dialysis or other renal replacement therapy (RRT) is required. Despite the advent of newer drugs, more sophisticated RRT equipment, and increased awareness of the problem, little has changed relative to patient outcomes, which remain poor. Similarly, limited options exist in patients with known risk factors for AKI to prevent its development due to iatrogenic causes (e.g., major surgery, exposure to contrast media).

Targeted Renal Therapy allows for direct delivery of therapeutically relevant doses of various pharmacological agents directly to the renal bed, potentially reducing dose limiting side effects of traditional IV therapy. With Targeted Renal Therapy, or TRT, the kidney can metabolize, conjugate, and/or clear a substantial portion of many agents immediately (known as the "renal first-pass" effect), reducing the amount that is returned to the systemic circulation via the renal veins, thus potentially reducing untoward side effects. While the existence of a renal first-pass effect has been hypothesized in the medical literature for some time, it has not been possible to take clinical advantage of this important physiological function prior to the advent of AngioDynamics' TRT. Thus, TRT has the potential to offer an additional preventative or treatment opportunity in those patients at risk for AKI, or with established AKI, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Physician-determined need for Benephit device/Targeted Renal Therapy
* Age >=18 years
* Ability to provide written informed consent

Exclusion Criteria:

* Patients who are participating in another IRB approved research study that precludes simultaneous enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For use in patients undergoing medical, interventional, or surgical procedures, where the procedure carries an elevated risk of iatrogenic acute kidney injury for the patient. Also indicated in patients who have demonstrated symptoms of acute kidney injury, and in whom arterial catheterization with the Benephit infusion systems is feasible.
Sampling Method: Non-Probability Sample
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Baptist Cardiac & Vascular Institute, Miami, Florida
  - HealthwoRx South Florida Research Solutions, Miramar, Florida
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - Cardiology Associates of NW Indiana, Munster, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - King's Daughters Medical Center, Ashland, Kentucky
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Sahetya Medical Institute, Bowling Green, Kentucky
  - Western Kentucky Heart and Lung, Bowling Green, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - St. John Hospital & Medical Center, Detroit, Michigan
  - St. Joseph Health Center, Saint Charles, Missouri
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Utah Cardiology PC, Layton, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia